CLINICAL TRIAL: NCT01111812
Title: Prediction of Weight Gain by Children and Adolescents That Participate in a Multi-disciplinary Intervention Program for Treatment of Overweight and Obese
Brief Title: Prediction of Weight Gain by Children and Adolescents
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Dan Nemet, MD, MD Prof., Meir Medical Center
Other Study IDs: MMC131-09CTIL
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Overweight; Obesity
Keywords: overweight; obese; children; weighing; weight
MeSH Terms: conditions — Overweight; Obesity; Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- weight measurements: This study include 1000 weight measurements of children and adolescence, boys and girls, ages 5-18, that taking pat in a multi-disciplinary intervention program for treatment of the overweight and obese in Meir medical center.

SUMMARY:
The 'Meir children's sport and health center' runs a multi-disciplinary intervention program for the treatment of overweight and obese children and adolescents. The program includes physical activity, dietary guidelines, medical supervision and behavioral treatment. The participants are routinely weighed once a week, at the same day and time, in order to supervise their progress. According to our experience, the child can predict his weight change, based on his "behavior" in the previous week. To our knowledge the overweight/obese child's ability to predict his weekly weight change, while participating in a multi-disciplinary intervention program, has never been tested.

DETAILED DESCRIPTION:
The aim of this study is to examine whether a child participating in a multi-disciplinary intervention program for treatment of the overweight and obese in Meir medical center, can predict his weight change during intervention before the actual weighing.

This study will include 1000 weight measurements of children and adolescents, boys and girls, ages 5-18 years. A patient might be measured several times.

The data will be collected during 6 mounts. in this period the program participants will be asked, discretely, before being weighed if, in there opinion, they had lost or gained weight in the past week, and how mach and why.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obese children and adolescence
* Boys and girls
* Ages 5-18
* That taking pat in a multi-disciplinary intervention program for treatment of the overweight and obese in Meir medical center

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: overweight and obese children and adolescence, boys and girls, ages 5-18
Sampling Method: Non-Probability Sample
Enrollment: 530 (Actual)
Dates: Start 2011-01; Primary Completion 2017-06 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Participants will be able to predict their weight change | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- 'Meir children's sport and health center', Kfar Saba, Israel